CLINICAL TRIAL: NCT07278817
Title: Study on the Monitoring of Traditional Chinese and Western Medicine Characteristics and Rehabilitation Program for ICIAM：A Cohort Study
Brief Title: Monitoring and Rehabilitation for ICIACI Rehabilitation：A Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Weifang Hospital of Traditional Chinese Medicine (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Jingyi Ren, Professor of medicine(Cardiology), Deputy Director of the Cardiology Department and Director of the Heart Failure Center, China-Japan Friendship Hospital
Other Study IDs: 2023ZD0502805-01
Record Dates: First submitted 2025-11-30; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Immune Checkpoint Inhibitor-Related Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICIACI-Rehab Cohort

SUMMARY:
Immune checkpoint inhibitor-associated cardiac injury (ICIACI) is a low-incidence but highly fatal adverse event. A significant knowledge gap exists regarding the disease characteristics and recovery status of patients during the ICIACI convalescent phase. The objectives of this study are to establish a national, multicenter cohort for this patient population and to comprehensively describe their clinical profiles from an integrated Traditional Chinese and Western medicine standpoint, as well as their current rehabilitation status.

DETAILED DESCRIPTION:
The cohort study consists of a retrospective and a prospective cohort, enrolling eligible rehabilitation ICIACI patients from multiple centers across China. The retrospective cohort records baseline assessment data from electronic medical records and clinical sources, including demographics, cancer diagnosis and immunotherapy details, laboratory tests, electrocardiograms, imaging studies, quality of life and exercise tolerance assessments, TCM syndrome scores, and rehabilitation information, to define TCM and Western medicine clinical characteristics and rehabilitation status. The prospective cohort patients are followed up at 2, 4, and 12 weeks after enrollment, with MACE as the primary endpoint and quality of life scores as the secondary endpoint, to evaluate influencing factors of rehabilitation and its impact on prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years, inclusive
* Malignancy confirmed by cytology or histopathology
* Diagnosis of ICIACI following ICI therapy
* Assessed by the Multidisciplinary Team for Immune-Related Adverse Events as clinically recovered and entering the rehabilitation.

Exclusion Criteria:

* Diagnosis of fulminant myocarditis or cardiac function of NYHA IV
* Clear evidence suggesting cardiac injury not attributable to ICIs
* Concurrent acute cardiovascular events or malignant arrhythmias
* Coexisting severe immune-related adverse events affecting other organ systems
* Associated severe systemic diseases, such as severe hepatic or renal insufficiency, or severe infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Under the established protocol, patients presenting with ICIACI will be enrolled from the China-Japan Friendship Hospital, Fuwai Hospital of the Chinese Academy of Medical Sciences, the Second Affiliated Hospital of Nanchang University, and Weifang Hospital of Traditional Chinese Medicine during the period from December 2025 to July 2028.
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 2, 4, and 12 weeks after enrollment
  Cardiovascular Death, Cardiac Arrest, Cardiogenic Shock, High-Grade Atrioventricular Block

SECONDARY OUTCOMES:
EQ-5D | 2, 4, and 12 weeks after enrollment
  This study employed the EuroQol 5-Dimensions 5-Level questionnaire (EQ-5D-5L). It consists of two parts:
  Health Description System:Responses were converted to a single health utility index score using the Chinese value set (range: -0.391 to 1.000). A higher score indicates better health-related quality of life.
  Visual Analogue Scale (EQ-VAS): Patients rated their current overall health from 0 (worst imaginable) to 100 (best imaginable). A higher score reflects better self-rated health.
  Changes in both the index score and EQ-VAS score from before to after the intervention were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Ren, Professor, Principal Investigator — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: No